CLINICAL TRIAL: NCT00120887
Title: Lupus Atherosclerosis Prevention Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Lupus Research Alliance (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: LAPS
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2006-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Atherosclerosis, SLE, statins
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Atherosclerosis | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
Cardiovascular disease, specifically from atherosclerosis, is the major cause of mortality in systemic lupus erythematosus (SLE) in developed countries. Coronary artery disease and stroke contribute to long-term morbidity in surviving patients. Atherosclerosis in SLE is multifactorial, with immune/inflammatory endothelial damage, traditional cardiovascular risk factors, and prothrombotic factors all playing important roles. Multiple groups have shown that hyperlipidemia is predictive of later atherosclerosis in SLE. In the general population, statins have become the drug of choice in preventing atherosclerotic events, through two mechanisms: lipid lowering that helps to prevent progression, and stabilization of plaques to prevent rupture. In the Lupus Atherosclerosis Prevention Trial we will determine if atorvastatin reduces the progression of atherosclerosis on helical computed tomography (CT) and carotid duplex. Recent work has confirmed that statins have an immunomodulatory role. This study will also determine whether statins improve clinical lupus activity or lupus serologies (anti-dsDNA and complement).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of SLE, confirmed by a faculty rheumatologist at Johns Hopkins.
* Patients must be 18 years of age or older
* Give informed consent.

Exclusion Criteria:

* SLE patients with a known atherosclerotic event, such as angina, myocardial infarction, or stroke, with an abnormal lipid profile for which a statin would be standard of care, are excluded.
* Pregnant patients (or patients planning to become pregnant in the next two years) are excluded.
* Patients who have known chronic liver disease, have unexplained elevation of their liver enzymes greater than 2 times the upper limit of normal , or an elevated CPK greater than 1.5 times the upper limit of the normal value for the patient's racial group, are excluded.
* Patients with triglycerides greater than 500 mg/dl or LDL greater than 190 in the absence of 2 risk factors (and who are unwilling to participate in a formal nutritional/lifestyle modification program that we recommend for them) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-04; Study Completion 2005-12

PRIMARY OUTCOMES:
This clinical trial of atorvastatin 40 mg vs. placebo will determine if atorvastatin will:. Reduce progression of atherosclerosis on helical CT or carotid duplex.
Determine whether atorvastatin 40 mg is more effective than placebo in retarding coronary calcification on multislice helical CT over two years.
Determine whether atorvastatin 40 mg is more effective than placebo in preventing new or preventing progression of old atherosclerotic plaque on carotid duplex over two years.
Determine whether atorvastatin 40 mg is more effective than placebo in preventing carotid intimal medial thickness on carotid duplex over two years.

SECONDARY OUTCOMES:
Determine whether a statin has an immunomodulatory benefit on SLE disease activity.
Determine whether there is a difference between atorvastatin and placebo arms in bone mineral density at one year, due either to improvement in, or prevention of, osteoporosis in the atorvastatin arm, or to progression in the placebo arm.
Determine predictors of atherosclerosis in SLE, including: a) cardiovascular risk factors; b) measures of SLE activity, damage and health status; c) antiphospholipid antibodies; d) renal function; e) treatment; and f) sociodemographic variables.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Petri, M.D.,MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Lupus Center 1830 E Monument Street, Ste 7500, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Petri MA, Kiani AN, Post W, Christopher-Stine L, Magder LS. Lupus Atherosclerosis Prevention Study (LAPS). Ann Rheum Dis. 2011 May;70(5):760-5. doi: 10.1136/ard.2010.136762. Epub 2010 Dec 21. PMID 21177297